CLINICAL TRIAL: NCT02125409
Title: Acetylsalicylic Acid and Colorectal Cancer Prevention: Exploring the Platelet Function of Its Mechanism of Action.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aragon Institute of Health Sciences (Other)
Collaborators: G. d'Annunzio University (Other); Catholic University, Italy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: D-13-01; 2013-004269-15 (EudraCT Number)
Record Dates: First submitted 2014-04-25; First posted 2014-04-29 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-05

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Group 1, individuals will be treated with ASA for 1 week; then blood and tissue samples (during the screening colonoscopy) will be collected at from 6-7 h after the last dose of ASA.
  Interventions: Drug: Acetylsalicylic acid; Procedure: Screening colonoscopy
- Group 2 (Experimental): Group 2, individuals will be treated with ASA for 1 week; then blood and tissue samples (during the screening colonoscopy) will be collected at 24 hours after the last dose.
  Interventions: Drug: Acetylsalicylic acid; Procedure: Screening colonoscopy

INTERVENTIONS:
Drug: Acetylsalicylic acid — One tablet of Adiro 100 mg will be administered daily for 7 days.
  Other Names: Adiro 100; ASA
Procedure: Screening colonoscopy

SUMMARY:
In a preliminary study in healthy subjects, the investigators determined the pharmacokinetic and pharmacodynamic of enteric-coated acetylsalicylic acid (ASA) (Adiro 100 mg, Bayer), and the variability (coefficient of variation), accuracy and precision of a novel biomarker of ASA action, i.e., quantification of the extent of COX-1 acetylation at serine-529, using a stable isotope dilution liquid chromatography multiple reaction monitoring/mass spectrometry (LC-MS) technique.

Now, the investigators will perform a clinical study in individuals undergoing Colorectal cancer (CRC) to validate the hypothesis that that low-dose ASA given once daily is acting primarily by selectively acetylating platelet COX-1 and suppressing its activity throughout the 24-hour dosing interval. In contrast, it is expected that the inhibitory effect on extra-platelet sources of COX-1 will be short-lasting, if any, affecting only partially COX-1, and this effect will be completely reversed at 24 hours after dosing. This is an important point which will strengthen the platelet hypothesis underpinning the apparent adequacy of a 24-hour dosing interval of ASA administration for the anticancer effect detected in cardiovascular trials.

These patients will be stratified into individuals with adenomas/carcinomas (20 to 30%) and patients without clinically detected adenomas/carcinomas (about 70 to 80%).

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, aged ≥ 18 and ≤ 69.
2. Patients should have an indication for screening colonoscopy

   1. First degree relative of patient with CRC.
   2. Personal history of adenomas.
   3. People older than 50 and FOBT positive
3. Routine hematological and biochemical parameters within the normal range.

Exclusion Criteria:

1. Allergy to ASA or other NSAIDs.
2. Previous use of ASA, NSAIDS, antiplatelet agents, corticosteroids or misoprostol in the previous 15 days and/or anticipated need for these drugs during the study period.
3. Peptic ulcer history or any other gastrointestinal disease that could be considered a contraindication for ASA use without the concomitant use of a proton-pump inhibitor.
4. Subjects with coagulation disorder or serious comorbid condition.
5. Malignancies, excluding CRC, diagnosed in the previous 5 years
6. Cigarette smoking, history of drug or alcohol abuse
7. Pregnant women or breast feeding

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Assessment of the degree of COX-1 acetylation by ASA administered for 1 week. | 7 hours after the 7th daily dose (group 1) and 24 hours after the 7th daily dose (group 2)
  It will be performed in platelets versus biopsies of the recto-colonic tissues.

SECONDARY OUTCOMES:
Changes from baseline in different biomarkers. | pre-drug on day 0 and after the 7th daily dose (6 hours for Group 1 and 24 hours for Group 2)
  It will be used a combining technique of liquid chromatography with mass spectrometry (LC-MS/MS) to quantify the level of acetylation of COX-1 in circulating platelets in subjects treated with ASA.
  Parameters of the composite measure:
  * haemochrome, AST, ALT, gamma-GT, alkaline phosphatase (AP), total bilirubin, total protein, glucose, creatinine, N, Na, K, Ca.
  * urine analysis: pH, protein, albumin, glucose, RBC, bilirubin, nitrites, leucocytes and sediment.
Changes from baseline in eicosanoid generation in vivo by measuring urinary metabolites derived from COXs. | pre-drug on day 0 and after the 7th daily dose (6 hours for Group 1 and 24 hours for Group 2)
  It will be performed by ultra-performance liquid chromatography tandem mass spectrometry-mass spectrometry (UPLC/MS/MS).
Changes in baseline platelet COX-1 | pre-drug on day 0 and after the 7th daily dose (6 hours for Group 1 and 24 hours for Group 2)
  By using human whole blood assay (serum TXB2) ex vivo
Change from baseline in plasma proteins of markers of angiogenesis. | pre-drug on day 0 and after the 7th daily dose (6 hours for Group 1 and 24 hours for Group 2)
  In blood sample by using an antibody array kit and Sphingosine-1 Phosphate (S1P) by immunoassay.
Assessment of ASA plasma levels. | pre-drug on day 0 and after the 7th daily dose (6 hours for Group 1 and 24 hours for Group 2)
  Will be performed whole blood aggregation test.
Changes from baseline of proteomic profile of selected angiogenesis factors, ie VEGF, FGF2, TGFbeta, EGF, PDGF, MMP, angiogenin, and angiogenesis inhibitors, ie endostatin, PF4, thrombospondin 1, alpha-macroglobulin, PAI 1 and angiostatin. | pre-drug on day 0 and after the 7th daily dose (6 hours for Group 1 and 24 hours for Group 2)
  It will be done in isolated platelets by using an antibody array kit and Sphingosine-1 Phosphate (S1P) by immunoassay.
Change from baseline in eicosanoid biosynthesis and protein expression of markers of growth and progression of colorectal cancer (such as COX-2, NF-Kb and PI3K/Akt/mTOR pathway). | pre-drug on day 0 and after the 7th daily dose (6 hours for Group 1 and 24 hours for Group 2)
  It will be done in normal tissues or pathological recto-colonic tissues.

CONTACTS AND LOCATIONS:
Overall Officials: Angel Lanas Arbeloa, Physician, Principal Investigator — Digestive disease service of Hospital Clinico Lozano Blesa
Locations (1):
- Hospital Clínico Universitario Lozano Blesa, Zaragoza, Zaragoza, Spain